CLINICAL TRIAL: NCT02164422
Title: Does Guanfacine Attenuate Stress-Induced Drinking?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Sherry McKee, Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1308012557; R01AA022285 (NIH)
Record Dates: First submitted 2014-05-23; First posted 2014-06-16 (Estimated); Results first posted 2021-04-21 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Alcohol Drinking
Keywords: Alcohol; Drinkers; Guanfacine
MeSH Terms: conditions — Alcohol Drinking | interventions — Guanfacine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Guanfacine 3mg/day (Experimental): Guanfacine 3mg/day
  Interventions: Drug: Guanfacine 3mg/day
- Guanfacine 1.5mg/day (Experimental): Guanfacine 1.5mg/day
  Interventions: Drug: Guanfacine 1.5mg/day
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Guanfacine 3mg/day — 3 mg/day Guanfacine with 3-week lead-in period. Maintained at steady state throughout lab sessions. After lab sessions, given taper supply of medication. Follow up 2 weeks after completion of taper.
  Other Names: Tenex
  Arms: Guanfacine 3mg/day
Drug: Guanfacine 1.5mg/day — 1.5 mg/day Guanfacine with 3-week lead-in period. Maintained at steady state throughout lab sessions. After lab sessions, given taper supply of medication. Follow up 2 weeks after completion of taper.
  Other Names: Tenex
  Arms: Guanfacine 1.5mg/day
Drug: Placebo
  Arms: Placebo

SUMMARY:
Evaluating the effect of guanfacine on alcohol consumption. The investigators hypothesize that guanfacine versus placebo will decrease the amount of alcohol consumption (mls consumed) during the 2-hour self-administration period across two laboratory sessions.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-65
* Able to read and write English
* Meets Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria for current (past 6 months) alcohol abuse or alcohol dependence

Exclusion Criteria:

* Participants with any significant current medical conditions, seizures, delirium or hallucinations, or other unstable medical conditions including HIV
* Current DSM-IV abuse or dependence on substances, other than alcohol abuse, alcohol dependence, or nicotine dependence
* Women who are pregnant or nursing
* Suicidal, homicidal or evidence of current (past 6-month) mental illness
* Meet DSM-IV criteria for current (past-6 month) attention deficit hyperactivity disorder (ADHD)
* Specific exclusions for administration of guanfacine not already specified include: EKG evidence at baseline screening of any clinically significant conduction abnormalities or arrhythmias; known intolerance for guanfacine or any alpha blocker; history of fainting, syncopal attacks, heart failure or myocardial infarction, or impaired liver as indicated by aspartate aminotransferase (AST), alanine aminotransferase (ALT) > 3x normal or renal function (estimated creatinine clearance <60 cc/min); treatment with any antihypertensive drug or any alpha-adrenergic blocker; use of any central nervous system (CNS) depressant (e.g., phenothiazines, barbiturates, benzodiazepines)
* Subjects likely to exhibit clinically significant alcohol withdrawal during the study.
* Individuals who are seeking treatment for drinking

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry A McKee, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Center for Clinical Investigations, Yale University, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Guanfacine 3mg/Day | Guanfacine 1.5mg/Day | Placebo
Started | 25 | 22 | 23
Completed | 24 | 20 | 23
Not Completed | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Guanfacine 3mg/Day | Guanfacine 1.5mg/Day | Placebo | Total
Number analyzed (Participants) | 24 | 20 | 23 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.21 (12.504) | 28.65 (10.594) | 37.04 (13.482) | 34.60 (12.754)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 8 | 20
  Male | 19 | 13 | 15 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 13 | 11 | 11 | 35
  White | 11 | 9 | 11 | 31
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 20 | 23 | 67

OUTCOME MEASURES:

1. Primary Outcome: mL Per 15 Minutes
Description: mL per 15 minutes during 2-hour ad-lib drinking period
Time Frame: 2 hour self administration period during lab sessions held on days 22 and 25
Measure: Mean (Standard Error); unit: mls of alcohol consumed per 15 minutes
Arm/Group | Guanfacine 3mg/Day | Guanfacine 1.5mg/Day | Placebo
Number analyzed (Participants) | 24 | 20 | 23
mls of alcohol consumed per 15 minutes | 85.850 (5.217) | 80.575 (5.567) | 114.104 (5.268)

ADVERSE EVENTS:
Time Frame: Day 1 to Day 22
Description: Treatment emergent adverse events
Arm/Group | Guanfacine 3mg/Day | Guanfacine 1.5mg/Day | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 3/25 | 2/22 | 3/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Guanfacine 3mg/Day (N=25) | Guanfacine 1.5mg/Day (N=22) | Placebo (N=23)
somnolence (General disorders) | 0 (0) | 0 (0) | 1 (1)
fatigue (General disorders) | 1 (1) | 0 (0) | 2 (2)
dizziness (General disorders) | 1 (1) | 0 (0) | 0 (0)
dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-21): https://cdn.clinicaltrials.gov/large-docs/22/NCT02164422/Prot_SAP_000.pdf